CLINICAL TRIAL: NCT04308603
Title: Multicentric Prospective Study to Screen Inborn Errors of Metabolism in Non-immune Hydrops Fetalis by Massively Parallel Sequencing
Brief Title: Multicentric Prospective Study to Screen Inborn Errors of Metabolism in Non-immune Hydrops (NIH) Fetalis by Massively Parallel Sequencing
Acronym: ANAMETAB-PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL19_0501; 2019-A02338-49 (Other: ID-RCB)
Record Dates: First submitted 2020-02-28; First posted 2020-03-16 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Non-Immune Hydrops Fetalis
Keywords: Non-immune hydrops fetalis; Multicentric prospective study; Next Generation Sequencing; Panel
MeSH Terms: conditions — Hydrops Fetalis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- pregnant patient whose fetuses have an antenatal NIH (Experimental): All pregnant patients whose fetuses have an antenatal revelation of NIH from the first trimester ultrasound scan will be included in this study.
  Interventions: Diagnostic Test: NON-IMMUNE HYDROPS FETALIS diagnosis

INTERVENTIONS:
Diagnostic Test: NON-IMMUNE HYDROPS FETALIS diagnosis — Amniotic liquid of each selected patients will be tested by both technic to describe and detect etiological information. Each patient will be tested using the current procedure with a defined panel of genes as well as with the NGS procedure. The results of both procedures will be compared.

SUMMARY:
A fetal hydrops, also called a fetal anasarca, is the buildup of fluid in the serosa and / or fetal subcutaneous tissue. The diagnosis is made by ultrasound, possibly from the first trimester of pregnancy.

The etiologies of hydrops can be immune or non-immune. The historically classic immune causes are linked to fetal-maternal alloimmunizations in erythrocyte blood groups. The implementation of systematic prevention of these anti rhesus immunizations since the 1970s has significantly reduced the incidence of immune hydrops Non-immune hydrops (NIH) now represent 90% of fetal hydrops. Known causes of NIH can be classified in several ways depending on the mechanism or organ involved.

The prognosis for NIH is closely linked to the cause. Fetal anemia due to maternal-fetal infections can heal spontaneously or give rise to in utero transfusions. Cardiac rhythm abnormalities are accessible to medical treatment. Chylothorax compressions may benefit from in utero drainage, but chromosomal or metabolic causes cannot benefit from antenatal care. The term of pregnancy in which the hydrops is discovered also has an impact on survival, which however remains poor.

In France, certain pathologies can be considered as particularly serious without the possibility of treatment and give rise to a request for medical termination of pregnancy. This possibility is subject to acceptance by two practitioners who are members of a multidisciplinary prenatal diagnostic center (CPDPN). This preliminary multidisciplinary reflection participates in the development of prenatal counseling with the greatest precision in diagnostic hypotheses. This prenatal advice is essential for a couple on the decision to make a pregnancy in progress but also for future pregnancies, given the 25% risk of recurrence due to the autosomal recessive mode of transmission.

Thus the current screening strategy for inherited metabolic diseases on amniotic fluid is fragmented. The resulting subdiagnosis explains the objective of the study of using the new high throughput sequencing techniques (NGS) in this indication. This approach should make it possible to reduce the number of cases classified as idiopathic, to allow the parents concerned to receive suitable genetic counseling with a view to new pregnancies, and to refine the knowledge of the prenatal epidemiology of these pathologies.

ELIGIBILITY:
Inclusion Criteria:

* patient> 18 years old
* Single Pregnancy
* Progressive pregnancy greater than 11 weeks: Fetal death in utero in a fetus previously known to be a carrier of non Immun Hydrops (NIH) is not an exclusion criterion.
* Presence of an ultrasound defined as follows and confirmed by a multidisciplinary prenatal diagnostic center CPDPN:
* Before 14 weeks: Generalized subcutaneous edema descending to the abdomen, associated or not with peri-visceral effusion
* After 14 weeks: presence of at least 2 of the following criteria: ascites, pleural effusion, pericardial effusion, subcutaneous edema, placental edema, hydramnios.
* Persistent hygroma after 14 weeks of amenorrhea
* Persistent isolated perivisceral effusions without etiologies found
* Patient having an invasive diagnostic sample (amniocentesis)
* Social insured in France
* Patient who signed the informed consent of the study

Exclusion Criteria:

* NIH whose diagnosis is known and confirmed as non-metabolic by a CPDPN
* Non-progressive pregnancy with Fetal Death in utero with normal previous ultrasound monitoring
* Refusal of invasive diagnostic sampling
* Patient under legal protection measure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Proportion of fetuses for which a genetic anomaly responsible for antenatal revelation Non Immun Hydrops by Next Generation Sequencing (NGS) analysis | during pregnancy after the 14th week of amenorrhea
  Proportion of fetuses for which a genetic anomaly responsible for antenatal revelation Non Immun Hydrops can be detected by Next Generation Sequencing (NGS) analysis of the gene panel incriminated in inherited metabolic malformation compared to the proportion of fetuses for which a genetic anomaly has been identified by the technique current standard biochemical.

SECONDARY OUTCOMES:
Comparison of percentage of etiology detected between the NGS technique and the biochemical technique. | during pregnancy after the 14th week of amenorrhea
  The percentage of the following etiology of interest (Cardiovascular abnormalities, Chromosomal abnormalities, Haematological abnormalities, infections, Thoracic anomalies, Twin-to-twin transfusion syndromes, Uro-Nephrological Anomalies, Abdominal anomalies, Lymphatic dysplasia, Fetal or placental tumors, osteochondrodysplasias. syndromic, Hereditary Metabolism Diseases) will be assessed and compared between the 2 methods.
time to return the results in days of NGS techniques | during pregnancy after the 14th week of amenorrhea
  The delay of answer will be defined by the time to return the results by analysis of the panel of genes tested compared to the current standard biochemical technique, measured between the date of completion of the prenatal diagnosis procedure and the date of communication of the results to the parents.
number of technical failure of these new tools of NGS techniques | during pregnancy after the 14th week of amenorrhea
  Number of technical failures: unable to extract DNA, too little DNA, failed sequencing), and analysis of these failures will be measured and compared to the current standard biochemical technique.
Number of cases where the interpretation of the genetic variants did not lead to a conclusion | during pregnancy after the 14th week of amenorrhea
  by the number of cases where the interpretation of the genetic variants highlighted did not allow concluding on the imputability for the clinical picture will be assessed of these new tools of NGS techniques
number of week of amenorrhea of gestation | immediately after the child birth
  number of week of amenorrhea of gestation will be measured
issue of the pregnancy | immediately after the child birth
  The percentage of death in utero, the percentage of medical termination of pregnancy, the percentage of neonatal survival and the percentage of pregnancy continued until the end will be calculated

CONTACTS AND LOCATIONS:
Locations (17):
- France (17):
  - CHU Besançon, Besançon
  - CHU Pellegrin, Bordeaux
  - Hôpital Femme Mère Enfant, Bron
  - Hôpital d'Estaing, Clermont-Ferrand
  - Hôpital Le Bocage, Dijon
  - CHU Grenoble, La Tronche
  - CHU Limoges, Limoges
  - Hopital Croix Rousse, Lyon
  - Hopital Nord, Marseille
  - CHU Marseille Timone, Marseille
  - CHU Montpellier, Montpellier
  - Hôpital Archet 2, Nice
  - APHP Trousseau, Paris
  - Hopital Lyon Sud, Pierre-Bénite
  - CHU Saint Etienne, Saint-Priest-en-Jarez
  - Hôpital Paule de Viguier;, Toulouse
  - CHU de Nancy Brabois,, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No